CLINICAL TRIAL: NCT04043065
Title: A Leap to Understand Glucoregulatory Effects of Liver-enriched Antimicrobial Peptide 2 (LEAP-2)
Brief Title: Liver-enriched Antimicrobial Peptide 2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Gubra ApS (Unknown)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, head of department, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LEAP-2
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study is designed as a clinical, placebo-controlled, double-blinded cross-over study involving two experimental study days.
Who Masked: Participant, Investigator
Masking Description: Day A and B will be conducted in a randomised, double-blinded order (blinded for the participant and the investigator) and noted by a third person not participating in the collection or analyses of data. The infusion order will be opened after the primary data analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEAP-2 (Experimental): Liver-enriched antimicrobial peptide 2
  Interventions: Biological: Liver-enriched antimicrobial peptide 2
- Placebo (Placebo Comparator): Saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Liver-enriched antimicrobial peptide 2 — Infusion of LEAP-2 during a 180 min grated glucose infusion.
  Arms: LEAP-2
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
The investigators aim to investigate the physiological importance of LEAP-2 in healthy volunteers focusing on its potential insulinotropic effects.

DETAILED DESCRIPTION:
The dramatic and almost immediate effects of Roux-en-Y gastric bypass (RYGB) surgery on type 2 diabetes (T2D) can only in part be explained by alterations in the plasma concentrations of known peptides. Thus, other - yet unknown - signals or hormones elicited from the endocrine cells of the small intestine may play an important role for the remission of T2D observed following RYGB. In a recent study, a predicted sequence of liver-enriched antimicrobial peptide 2 (LEAP-2) was shown to induce a glucose-stimulated insulin secretion in isolated human pancreatic islets. The fragment was subsequently identified to be circulating in human plasma in concentrations comparable to the circulating levels of other known gut secreted hormones, hereby validating that LEAP-2 is an endogenous circulating peptide.

The investigators hypothesise that LEAP-2 increases insulin secretion during a graded glucose infusion as assessed by plasma insulin and C-peptide compared with saline (placebo) in healthy subjects. The study is designed as a clinical, placebo-controlled, double-blinded cross-over study involving two experimental study days and ten young healthy male participants. The co-primary endpoints are the difference in plasma insulin levels during a graded glucose infusion and beta-cell secretion assessed by plasma C-peptide concentration relative to plasma glucose concentration between the two study days with either saline (placebo) or LEAP-2 infusion.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men
* Age between 18 and 25 years
* Body mass index between 20-25 kg/m2
* Informed consent

Exclusion Criteria:

* Anaemia (haemoglobin below normal range)
* ALAT and/or ASAT >2 times normal values or history of hepatobiliary and/or gastrointestinal disorder(s)
* Nephropathy (serum creatinine above normal range and/or albuminuria)
* Any physical or psychological condition that the investigator evaluates would interfere with trial participation including any acute or chronic illnesses
* Any ongoing medication that the investigator evaluates would interfere with trial participation.
* First- and second-degree relatives with diabetes
* Regular tobacco smoking

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Plasma insulin | -45 to 180 minutes
  Difference in plasma insulin levels
Beta-cell secretion | -45 to 180 minutes
  Beta-cell secretion assessed by plasma C-peptide concentration relative to plasma glucose concentration

SECONDARY OUTCOMES:
LEAP-2 | -45 to 210 minutes
  Plasma concentrations of LEAP-2
Resting energy expenditure | -20 to 160 minutes
  Changes in resting energy expenditure using indirect calorimetry
Appetite, satiety, and general well-being | -45 to 210 minutes
  Appetite, satiety, and general well-being assessed by visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Study Director — University Hospital, Gentofte, Copenhagen
Locations (1):
- Center for Clinical Metabolic Research, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No